CLINICAL TRIAL: NCT07220642
Title: Efficacy and Safety of Cagrilintide for Weight Management in Participants With Overweight or Obesity
Brief Title: Weight Loss in People Living With Overweight or Obesity Following Treatment With Cagrilintide
Acronym: RENEW 1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9833-8242; U1111-1314-8906 (Other: World Health Organization (WHO)); 2024-519530-24 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-10-23; First posted 2025-10-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — cagrilintide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cagrilintide (Experimental): Participants will receive cagrilintide subcutaneously once weekly for 64 weeks.
  Interventions: Drug: Cagrilintide
- Placebo (Placebo Comparator): Participants will receive placebo matched to cagrilintide subcutaneously once weekly for 64 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cagrilintide — Cagrilintide will be administered subcutaneously with a pen-injector as an adjunt to lifestyle intervention counselling.
  Arms: Cagrilintide
Drug: Placebo — Placebo matched to cagrilintide will be administered subcutaneously with a pen-injector as an adjunt to lifestyle intervention counselling.
  Arms: Placebo

SUMMARY:
This study will look at how much cagrilintide helps people with overweight or obesity lower their body weight. Cagrilintide is a new investigational medicine. Doctors may not yet prescribe cagrilintide. Participants will either get cagrilintide or placebo. Which treatment participants get is decided by chance. Participants are two times more likely to get cagrilintide than placebo. Like all medicines, the study medicine may have side effects. Possible side effects will be followed carefully during the study. For each participant, the study will last for about 1 year and 6 months.

ELIGIBILITY:
Inclusion criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study
* Female or male (sex at birth)
* Age 18 years or above at the time of signing the informed consent
* History of at least one self-reported unsuccessful dietary effort to lose body weight (a*)
* Body mass index (BMI) greater than or equal to >= 30.0 kilogram per square meter (kg/m^2), or BMI greater than or equal to >= 27.0 kg/m^2 with the presence of at least one weight related comorbidity including, but not limited to, hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease (a*)

Exclusion criteria:

* History of type 1 or type 2 diabetes (a*)
* Treatment, or intention to initiate treatment, with any medication prescribed for the indication of weight management within 180 days before screening (a*)
* Previous dosing of marketed or non-marketed amylin-based compounds (a*) (a*) - As declared by the participant, reported in the medical records or at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-05-26 (Estimated); Study Completion 2027-07-14 (Estimated)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 64)
  Measured as percentage (%) of body weight.
Number of participants with achievement of greater than or equals (>=) 5 percent (%) body weight reduction | From baseline (week 0) to end of treatment (week 64)
  Measured as count of participants.

SECONDARY OUTCOMES:
Number of participants with achievement of >= 10 % body weight reduction | From baseline (week 0) to end of treatment (week 64)
  Measured as count of participants.
Number of participants with achievement of >= 15 % body weight reduction | From baseline (week 0) to end of treatment (week 64)
  Measured as count of participants.
Change in waist circumference | From baseline (week 0) to end of treatment (week 64)
  Measured as centimeter (cm).
Ratio to baseline in triglycerides | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline in high sensitivity C-Reactive Protein (hsCRP) | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Change in Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function score | From baseline (week 0) to end of treatment (week 64)
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. The physical function score ranges from 0-100.
Change in body weight | From baseline (week 0) to end of treatment (week 64)
  Measured as kilogram (kg).
Change in SF-36v2® Health Survey Acute (SF-36v2® Acute) physical component summary score | From baseline (week 0) to end of treatment (week 64)
  Measured as score on a scale. SF-36v2 Acute measures Health-Related Quality of Life (HRQoL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 Acute scores are norm-based scores, that is. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Higher scores indicate better functional health and well-being. The physical component summary score ranges from 6.1 to 79.7.
Change in SF-36v2® mental component summary score | From baseline (week 0) to end of treatment (week 64)
  Measured as score on a scale. SF-36v2 Acute measures Health-Related Quality of Life (HRQoL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 Acute scores are norm-based scores, that is. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Higher scores indicate better functional health and well-being. The mental component summary score ranges from -3.8 to 78.7.
Change in IWQOL-Lite-CT total score | From baseline (week 0) to end of treatment (week 64)
  Measured as score on a scale. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. The total score ranges from 0-100.
Number of participants with achievement of at least 14.6-point increase in IWQOL-Lite-CT Physical Function score (yes/no) | From baseline (week 0) to end of treatment (week 64)
  Measured as count of participants. IWQOL-Lite-CT measures weight related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Higher scores indicate better levels of functioning. The physical function score ranges from 0-100.
Change in Systolic Blood Pressure (SBP) | From baseline (week 0) to end of treatment (week 64)
  Measured as millimeter of mercury (mmHg).
Change in Diastolic Blood Pressure (DBP) | From baseline (week 0) to end of treatment (week 64)
  Measured as mmHg.
Ratio to baseline of total cholesterol | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline of High-Density Lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline of Low-Density Lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline of Very Low-Density Lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline of non-HDL cholesterol | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Ratio to baseline of free fatty acids | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Change in glycated haemoglobin (HbA1c) percentage-points (%-points) | From baseline (week 0) to end of treatment (week 64)
  Measured as %-points.
Change in HbA1c millimoles per mole (mmol/mol) | From baseline (week 0) to end of treatment (week 64)
  Measured as mmol/mol.
Change in Fasting Plasma Glucose (FPG) millimoles per litre (mmol/L) | From baseline (week 0) to end of treatment (week 64)
  Measured as mmol/L.
Change in FPG milligrams per deciliter (mg/dL) | From baseline (week 0) to end of treatment (week 64)
  Measured as mg/dL.
Ratio to baseline in fasting serum insulin | From baseline (week 0) to end of treatment (week 64)
  Measured as ratio.
Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to end of study (week 71)
  Measured as count of events.
Number of treatment emergent serious adverse events (TESAEs) | From baseline (week 0) to end of study (week 71)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (40):
- United States (9):
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Univ of Colorado at Denver, Aurora, Colorado
  - Florida Inst For Clin Res LLC, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Walgreens - Store 11760, Oak Park, Illinois
  - Midwest Inst For Clin Res, Indianapolis, Indiana
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Selma Medical Associates, Winchester, Virginia
- Argentina (2):
  - CIPREC Pueyrredon, Buenos Aires
  - CEDIC Centro de Investigación Clínica, CABA
- Australia (2):
  - Sydney Cardiometabolic Centre, Liverpool, New South Wales
  - Hunter Diabetes Centre, Merewether, New South Wales
- Canada (8):
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - Hamilton Medical Rsrch Grp, Hamilton, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Milestone Research, London, Ontario
  - Centricity Research Oshawa, Oshawa, Ontario
  - Centricity Research Toronto, Toronto, Ontario
  - Centricity Research Mirabel, Mirabel, Quebec
- France (2):
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec, Saint-Herblain
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Germany (3):
  - InnoDiab Forschung GmbH, Essen
  - Wendisch - Dahl Hamburg - DZHW, Hamburg
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
- Italy (4):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCS, Rome, RM
  - AOUP Giaccone Palermo, Palermo, Sicily
  - A.O.U. Bologna_ Policlinico S.Orsola Malpighi, Bologna
  - IRCCS Ospedale San Raffaele Milano, Milan
- Norway (3):
  - Haukeland Universitetssykehus, Bergen
  - Drammen sykehus - Vestre Viken HF, Drammen
  - St. Olavs Hospital HF, Trondheim
- Poland (4):
  - Osteo-Medic s.c. A. Racewicz, J. Supronik, Bialystok
  - Care Clinic Sp. z o. o., Katowice
  - Terpa Sp. z o.o. Sp. k., Lublin
  - NBR Polska Tomasz Klodawski, Warsaw
- United Kingdom (3):
  - Oak Tree Surgery, Liskeard, Cornwall
  - North Coast Medical Ltd, Newquay, Cornwall
  - Brunel Medical Practice, Torquay, Devon

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com